CLINICAL TRIAL: NCT05585970
Title: Comparison of Procalcitonin Level in Normal Population and in Chronic Kidney Disease Patients Who Don't Have Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rofida Saadeldin Farghaly, resident doctor at CLINICAL PATHOLOGY department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-10-06
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Disease Patients Who Don't Have Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy Control individuals (Active Comparator)
  Interventions: Diagnostic Test: procalcitonin
- CKD patients (Active Comparator)
  Interventions: Diagnostic Test: procalcitonin
- ESRD on regular hemodialysis (Active Comparator)
  Interventions: Diagnostic Test: procalcitonin

INTERVENTIONS:
Diagnostic Test: procalcitonin — The PCT level in healthy individual without infection is below the limit of detection (0.01 ng/mL), and it is significantly elevated under the stimulation of pathogens
  Other Names: Kidney function tests . ESR. CRP. CBC

SUMMARY:
Chronic kidney disease (CKD) is a life threatening condition with high risk of pre-term death and need for dialysis. It is defined as kidney damage that has continued for more than 3 months as characterized by structural or functional abnormalities of the kidney, with or without decreased glomerular filtration rate (GFR). It is also defined as GFR < 60mL/min/1.73 m2 for more than 3 months, with or without structural kidney damage.

The PCT level in healthy individual without infection is below the limit of detection (0.01 ng/mL), and it is significantly elevated under the stimulation of pathogens. However, due to the pre-existing endogenous inflammation that occurs in CKD patients and the impaired kidney clearance, the reference range that applies to the general population may not be appropriate for diagnosing infections in CKD patients. More recently, debate has continued regarding whether the PCT level is increased in CKD patients without infection, and the optimal reference for CKD patients remains undetermined

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease patients.
* ESRD patients

Exclusion Criteria:

Any condition of infection or sepsis such as :

* Fever
* Increased TLC above normal
* Tachycardia
* Tachypnea
* Disturbed conscious level

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
procalcitonin Level | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosengren BI, Sagstad SJ, Karlsen TV, Wiig H. Isolation of interstitial fluid and demonstration of local proinflammatory cytokine production and increased absorptive gradient in chronic peritoneal dialysis. Am J Physiol Renal Physiol. 2013 Jan 15;304(2):F198-206. doi: 10.1152/ajprenal.00293.2012. Epub 2012 Nov 14. PMID 23152294
- [Background] Hamad A, Ismail H, Elsayed M, Kaddourah A, Ahmed H, Ibrahim R, Ali A, Alali F. The epidemiology of acute peritonitis in end-stage renal disease patients on peritoneal dialysis in Qatar: An 8-year follow-up study. Saudi J Kidney Dis Transpl. 2018 Jan-Feb;29(1):88-94. doi: 10.4103/1319-2442.225203. PMID 29456212
- [Background] Kim HJ, Vaziri ND. Contribution of impaired Nrf2-Keap1 pathway to oxidative stress and inflammation in chronic renal failure. Am J Physiol Renal Physiol. 2010 Mar;298(3):F662-71. doi: 10.1152/ajprenal.00421.2009. Epub 2009 Dec 9. PMID 20007347
- [Background] Chan YL, Tseng CP, Tsay PK, Chang SS, Chiu TF, Chen JC. Procalcitonin as a marker of bacterial infection in the emergency department: an observational study. Crit Care. 2004 Feb;8(1):R12-20. doi: 10.1186/cc2396. Epub 2003 Nov 20. PMID 14975050